CLINICAL TRIAL: NCT00322036
Title: Phase 3 Multinational, Randomized, Double Blind, Placebo Controlled Study of the Effect of Daily Treatment With MPC-7869 on Measures of Cognition, Activities of Daily Living and Global Function in Subjects With Mild Dementia of the Alzheimer's Type
Brief Title: Global Efficacy Study of MPC-7869 to Treat Patients With Alzheimer's
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Myriad has discontinued the development of Flurizan.
Sponsor: Myrexis Inc. (Industry)
Responsible Party: Ed Swabb, MD, Myriad Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MPC-7869-05-010.01
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Alzheimer Disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — tarenflurbil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Oral 800 mg BID dosing
  Interventions: Drug: MPC-7869
- 2 (Placebo Comparator): Oral BID dosing
  Interventions: Drug: MPC-7869

INTERVENTIONS:
Drug: MPC-7869 — Oral 800 mg BID
  Arms: 1
Drug: MPC-7869 — Oral BID dosing
  Arms: 2

SUMMARY:
This is a multinational, randomized, double blind, placebo controlled, parallel group study comparing the safety and efficacy of daily dosing of 800 mg twice daily MPC-7869 to placebo. Study subjects will have the diagnosis of mild dementia of the Alzheimer's type. Subjects may be taking approved medication for Alzheimer's disease provided the dose has been stable for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Have had a diagnosis of probable Alzheimer's disease
2. Men or women ages greater than or equal to 55 years and living in the community at the time of enrollment (ie, not living in a rest home or nursing care facility).
3. Signed the subject Informed Consent Form (ICF) and is willing and able to participate for the duration of the study.
4. Ability to read and understand English, Dutch, Danish, Flemish, French, German, Italian, Spanish or Swedish to ensure compliance with cognitive testing and study visit procedures.
5. At least 6 years of education, or sufficient work history to exclude mental retardation.
6. Female subjects must be surgically sterile or postmenopausal for > 1 year.
7. Adequate vision and hearing to participate in study assessments.
8. Subjects must have a reliable caregiver who can read, understand and speak same language.

Exclusion Criteria:

1. Current evidence of other causes of dementia.. .
2. History of, or evidence of, active malignancy, except for basal cell carcinoma or squamous cell carcinoma of the skin, within the 24 months prior to entry. Men with prostate cancer may be enrolled at the discretion of the sponsor.
3. Use of any investigational therapy within 30 days, or 5 half-lives, whichever is longer, and/or use of AD immunotherapy prior to screening.
4. Major surgery and related complications not resolved within 12 weeks prior to Day 1.
5. Previous participation in an MPC-7869 clinical study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2006-05; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Cognition and activities of daily living | 18 mos

SECONDARY OUTCOMES:
Global function and cognition | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Laughlin, MD, Study Director — Myrexis Inc.
Locations (92):
- United States (23):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Costa Mesa, California
  - San Diego, California
  - New Haven, Connecticut
  - Deerfield Beach, Florida
  - Delray Beach, Florida
  - Gainsville, Florida
  - Hollywood, Florida
  - Miami, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Boston, Massachusetts
  - Farmington Hills, Michigan
  - St Louis, Missouri
  - Rochester, New York
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Dallas, Texas
  - Salt Lake City, Utah
- Belgium (6):
  - Aalst
  - Antwerp
  - Edegem
  - Hasselt
  - Leuven
  - Sint-Truiden
- Canada (16):
  - Calgary, Alberta
  - Medicine Hat, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Moncton, New Brunswick
  - Saint John, New Brunswick
  - Halifax, Nova Scotia
  - Kingston, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Peterborough, Ontario
  - Toronto, Ontario
  - Greenfield Park, Quebec
  - Montreal, Quebec
  - Verdun, Quebec
  - Regina, Saskatchewan
- Denmark (2):
  - Odense
  - Odense C
- France (10):
  - Bordeaux
  - Dijon
  - Marseille
  - Montpellier
  - Nice
  - Reims
  - Rennes
  - Saint-Herblain
  - Toulouse
  - Tours
- Germany (12):
  - Berlin
  - Bochum
  - Bonn
  - Darmstadt
  - Düsseldorf
  - Freiburg im Breisgau
  - Hamburg
  - Heidelberg
  - Leipzig
  - Mannheim
  - München
  - Schwerin
- Italy (5):
  - Brescia
  - Milan
  - Perugia
  - Pisa
  - Roma
- Netherlands (3):
  - 's-Hertogenbosch
  - Amsterdam
  - Blaricum
- Spain (4):
  - Barcelona
  - Bilbao
  - Getafe. Madrid
  - Madrid
- Lund, Sweden
- Basel, Switzerland
- United Kingdom (9):
  - Bath, England
  - London, England
  - Oxford, England
  - Sheffield, England
  - Swindon, England
  - Belfast, Northern Ireland
  - Glasgow, Scotland
  - Penarth, Wales
  - Southhampton